CLINICAL TRIAL: NCT00900718
Title: Comparison of Straumann Bone Ceramic (SBC) and Bio-Oss in Combination With Guided Tissue Regeneration (GTR) for Volume Preservation of Alveolar Ridge After Tooth Extraction: a Randomised, Single Blind, Controlled Clinical Trial
Brief Title: Comparison of Straumann Bone Ceramic and Bio-Oss With Guided Tissue Regeneration for Alveolar Ridge Preservation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR 03/05
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Transplantation, Heterologous

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Straumann Bone Ceramic (Experimental): Bone augmentation, after tooth extraction, with Straumann Bone Ceramic (synthetic bone graft material) in combination with resorbable collagen membrane Bio-Gide.
  Interventions: Device: Straumann Bone Ceramic
- Bio-Oss (Active Comparator): Bone augmentation, after tooth extraction, with Bio-Oss (bovine-derived xenograft)in combination with resorbable collagen membrane Bio-Gide.
  Interventions: Device: Bio-Oss

INTERVENTIONS:
Device: Straumann Bone Ceramic — Bone augmentation, after tooth extraction, with Straumann Bone Ceramic (synthetic bone graft material) in combination with resorbable collagen membrane Bio-Gide.
  Other Names: Synthetic Bone Substitute
  Arms: Straumann Bone Ceramic
Device: Bio-Oss — Bone augmentation, after tooth extraction, with Bio-Oss (bovine-derived xenograft)in combination with resorbable collagen membrane Bio-Gide.
  Other Names: Xenograft
  Arms: Bio-Oss

SUMMARY:
The purpose of this study is to compare a new biomaterial with an already existing treatment principle (Bio-Oss/Bio-Gide) with regard to their ability to preserve the dimensions of the alveolar ridge and to promote bone regeneration and to evaluate the early survival rate of dental implants placed in the augmented socket area and to assess radiographically and clinically changes of peri-implant soft and hard tissues.

DETAILED DESCRIPTION:
This is prospective, randomized, single-blind, controlled, single center study. The total study duration for each patient should be 12 +/- 1 month.

In total 13 visits per patient are scheduled in this study.

The study devices Straumann Bone Ceramic and Bio-Oss are CE-marked, and approved by the FDA. The products are used within the indication.

One center in the Inited Kingdom will participate.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have voluntarily signed the informed consent
* Males and females, 18 years to 75 years of age
* Patient needs single tooth extraction in mandibular or maxillary incisor or pre-molar region and would benefit from prosthetic reconstruction with a dental implant
* Patients must be committed to the study and must sign informed consent
* Patient in good general health as documented by self assessment

Exclusion Criteria:

Systemic exclusion criteria

* Patient who has any known diseases (not including controlled diabetes mellitus), infections or recent surgical procedures within 30 days of study initiation
* Female patient who are pregnant or lactating or of child bearing potential not using acceptable methods of birth control (hormonal, barriers or abstinence
* Patient who are on chronic treatment (i.e., two weeks or more) with any medication known to affect oral status (e.g., phenytoin, dihydropyridine calcium antagonists, cyclosporine, and non-steroidal anti-inflammatory drugs) within one month of baseline visit
* Patient who are on concomitant anticoagulant therapy of warfarin (coumadine), clopidogrel, ticlopidine or once daily asprin of more than 81 mg.
* Patient who knowingly has HIV or Hepatitis
* Physical handicaps that would interfere with the ability to perform adequate oral hygiene
* Patient who has undergone administration of any investigational drug within 30 days of study initiation.
* Alcoholism or chronically drug abuse causing systemic compromisation
* Patient who is a heavy smoker (>10/cigarettes per day).
* Patient is suffering from a known psychological disorder
* Patient has limited mental capacity or language skills such that study information cannot be understood, informed consent cannot be obtained, or simple instructions cannot be followed

Local exclusion criteria

* Uncontrolled or untreated periodontal disease
* Bone defects that excludes implant restoration
* Patient who has a full mouth plaque level >30 % at the enrolment visit
* Mucosal diseases such as erosive lichen planus
* History of local radiation therapy
* Presence of oral lesions (such as ulceration, malignancy)
* Severe bruxing or clenching habits
* Persistent intraoral infection
* Patients presenting clinical and radiological signs and symptoms of maxillary sinus disease
* Patient presents an acute endodontic lesion in the test tooth or in the neighbouring areas to the experimental procedure (sites with presence of an asymptomatic chronic lesion are eligible)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-02; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The changes of bone level between baseline and 32 week post-extraction | baseline and 32 week post-extraction

SECONDARY OUTCOMES:
implant success and survival rate | 1 year post implant loading

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Donos, DDS, MS, PhD, Principal Investigator — Eastman Dental Institute
Locations (1):
- Eastman Dental Institute, University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No